CLINICAL TRIAL: NCT05286632
Title: Evaluation of Performance and Safety of App KidneYou, an Innovative Digital Therapy, in Improving Health of Patients with Chronic Kidney Disease (CKD) by Increasing Their Adherence to Dietary, Exercise Regimens or Mindfulness Program
Brief Title: KidneYou - Innovative Digital Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advice Pharma Group srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ADVICE-001-2022
Record Dates: First submitted 2022-02-25; First posted 2022-03-18 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Diseases; Diabetes; Arterial Hypertension; Chronic Glomerulonephritis; Cystic Kidney Diseases; Polycystic Kidney; Nephronophthisis; Cortical Cystic Disease; Cystic Diseases; Tuberous Sclerosis; Albuminuria; Treatment Adherence; Treatment Adherence and Compliance
Keywords: Digital Therapeutics; Digital Medicine; Adherence; Software; Software Medical Device; Quality of life; Digital Therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Hypertension; Kidney Diseases, Cystic; Polycystic Kidney Diseases; Nephronophthisis, familial juvenile; Tuberous Sclerosis; Albuminuria; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: This is an interventional, multicentric, randomized, double arm, comparative, parallel, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KidneYou APP (Experimental): In patients randomized in Group A (intervention group) the NP program will be administered by means of App KidneYou. Each patient will select the assigned daily menu or the proposed alternatives, following instructions reported for breakfast, mid-morning snack, lunch, afternoon snack, and dinner.
  Patients randomized to Group A (intervention group) will be administered the PA program by means of App KidneYou. Each patient will follow the assigned exercise program (i.e., recommended type of PA, minutes of exercise/day, number of days/week, level of intensity).
  Only patients randomized to Group A (KidneYou users) will be invited by the investigator to follow stress-reducing activities. This difference between the two groups is based on the nature of the mindfulness program, consisting solely of multimedia contents.
  Interventions: Device: KidneYou APP
- Standard of care control group (No Intervention): In patients randomized in Group B (control group) the NP program will be administered by means of a paper diary containing the entire range of daily menu and related alternatives needed to terminate the 3-month study period.
  Patients randomized to Group B (control group) will be administered the PA program by means of a paper diary containing the entire range of exercises needed to terminate the 3-month study period.
  The stress reduction program is not a "standard of care" currently used within the treatment strategy of CKD patients, neither through face-to-face visits with a specialist, nor through multimedia content.
  Patients provided with paper diary and randomized in Group B (KidneYou non-users) represent the population followed by the current "standard of care" and will not be provided with any multimedia content in the context of their participation in the present study.

INTERVENTIONS:
Device: KidneYou APP — KidneYou is a medical device designed to deliver digital therapy (DT) to patients. The DT utilizes high quality digital technologies to stimulate lifestyle changes in patients. KidneYou has been set up to improve the commitment of patients in following therapeutic directives (i.e. nutritional programs, daily/weekly physical activities) to manage their chronic diseases like CKD. Moreover, KidneYou can improve patient's awareness about his/her disease (mindfulness) so as to increase the individual human ability to be fully present at the ongoing disease's condition and react to it in active and positive manner. Particularly, the mindfulness program contained in this App has been designed to increase the patient's psychological and mental health, aiming at decreasing the perceived stress due to the underlying disease and to the attempts of life-style changes (i.e., healthy diet and physical activity) which may initially negatively affect the subject's natural attitudes.
  Arms: KidneYou APP

SUMMARY:
The aim of the study is to assess the improvement of health in patients affected by CKD when they are exposed to non-pharmacological treatment strategies as nutritional program (NP), physical activity program (PA) and mindfulness program (MP), when they are conveyed to the patient by means of digital technologies or not. In the present study, non-pharmacological interventions conveyed by a digital technology (investigational arm) will be compared to a standard, paper-based approach (control arm).

DETAILED DESCRIPTION:
KidneYou is a medical device designed to deliver digital therapy (DT) to patients. The DT, as part of Digital Health, utilizes high quality digital technologies to stimulate lifestyle changes in patients. KidneYou has been set up to improve the commitment of patients in following therapeutic directives (i.e. nutritional programs, daily/weekly physical activities) to manage their chronic diseases like CKD. Moreover, KidneYou can improve patient's awareness about his/her disease (mindfulness) so as to increase the individual human ability to be fully present at the ongoing disease's condition and react to it in active and positive manner.

The aim of this study is to determine whether the medical device KidneYou, randomly assigned to CKD patients (G3b/G4 categories; A1/A2 categories), can improve the CKD-related patient's health conditions by positive changes in the subject's lifestyle (i.e., healthy eating, physical activity participation) and by means of cumulative stress reduction (i.e., mindfulness program) originating from the underlying chronic disease and from diagnosis and treatment interventions necessary to manage it. Some lifestyle programs (i.e., nutrition and physical exercises) will be delivered to both randomized groups by different modalities (i.e. with/without KidneYou), while other programs (i.e., mindfulness) will only be accessible to KidneYou users, requiring a technology support for the multimedia content to be self-administered daily by the App. This innovative method avoids a daily face-to-face intervention administered by healthcare professionals for mental health treatments. Broadly speaking, it is expected that KidneYou may improve a patient's adherence to clinical advices and consequently patient's health condition in users compared to non-users. The enrolled subjects will be randomly assigned to one of the two treatment arms according to a parallel-group design. Subjects included in Group A (intervention group) will be provided with KidneYou, while patients in Group B (non-equivalent group) will be used as control. The study will enrol 210 subjects, both genders, aged ≥18 years, to obtain 190 overall valuable subjects (95 each group). The recruitment period will last 12 months.

For each patient the treatment will last 3 consecutive months (12 weeks) during which lifestyle changes will be implemented with/without KidneYou. At the end of this period the lifestyle program will be terminated, followed by a follow-up visit after 1 further month (16 weeks). The follow-up visit will be used to observe the sustained effects on patient's health 30 days after termination of the change lifestyle programs administered to patients with and without KidneYou.

At the beginning of the study, patients will be evaluated for their stress level by means of the Perceived Stress Scale (PSS) by Cohen (Cohen, 1983). Specifically, it will be used the Italian translation of PSS-10, which is a 10-item questionnaire designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. To customize the stress measurement to the population age range expected in this study, according to Norm Table for the PSS 10-item inventory, a cut-off of 12 points was chosen. Therefore, all subjects with a score >12 in the PSS questionnaire delivered at the first study visit (V0), will be considered to have a higher stress level above normal and to have one of the major inclusion criteria.

Each subject will undergo 4 (four) visits and will be examined according to the following schedule:

* V0 - Baseline
* V1 - 6 weeks after baseline (Day 42±2)
* V2 - 12 weeks after baseline (Day 84±2. End of lifestyle program administration)
* V3 - 4 weeks after V2 (Day 112±4. Follow-up visit and End of Study [EOS] visit)

Benefit/Risk Assessment Benefits for patients resulting from study implementation are the simultaneous application of the three non-pharmacological programs for improving the health of CKD patients. The expected results are that the simultaneous use of the three programs will allow greater improvements than those achieved so far with the separate use of programs. Instead of the experimental evidence published so far, the present study intends to measure the objective benefits rather than the perceived ones by CKD patients. For this, the composite primary objective/endpoint consists of easily measurable objective markers.

Improvements are expected in both treatment groups, as food and physical programs will also be implemented in the control (KidneYou non-users) group. However, in the investigational group (KidneYou users) it is assumed to achieve higher benefits, thanks to the possibility to offer, by means of the App software, the third psychological program (mindfulness) consisting of multimedia contents. The higher expected benefits in the investigational group are justified by the greater attractiveness of the App compared to paper diary in the control group, with a consequent increase in compliance and effectiveness in KidneYou users.

Possible risks that can be anticipated in this specific study population may be related to clinical events emerging from adherence to at least one of the three non-pharmacological programs, such as hypoglycemia, nausea, vomiting, gastrointestinal discomfort, physical accidents during exercises, hypertensive crises, obsessive feeling about exercise and food intake, anxiety/guilt when not reaching assigned exercise or food intake goals, interferences with subject's daily activities and/or social life, neuroses about individual body image or any other adverse experience.

Primary Objective

- To improve the quality and quantity of dietary intake in patients using KidneYou compared to patients unprovided with the App after 3 months of customized Nutritional Program (NP).

OR

- To increase energy expenditure in patients using KidneYou compared to patients unprovided with KidneYou after 3 months of customized Physical Activity Program (PA).

OR

- To relieve the stress related to the underlying CKD condition in patients using KidneYou compared to patients unprovided with KidneYou after 3 months of study.

Secondary Objectves

1. To help patients to achieve two or more of the above-mentioned objectives.
2. To describe each primary objective achieved in each randomized group.
3. To stratify the primary objective results by G3b and G4 category of CKD classification
4. To stratify the primary objective results by A1 and A2 category of CKD classification.
5. To assess the degree of azoturia reduction (g/24h) in each treatment group during the study.
6. To assess differences in azoturia reduction (g/24h) between the two randomized groups during the study.
7. To assess the degree of physical function improvements in each treatment group during the 6-MWT.
8. To assess differences in physical function improvements between the two randomized groups during the study.
9. To assess the degree of physical activity increase (minutes) in each treatment group during the study.
10. To assess the degree of stress reduction (Perceived Stress Scale [PSS] of Cohen) in each treatment group during the study.
11. To assess differences of stress reduction (Perceived Stress Scale [PSS] of Cohen) between the two randomized groups during the study.
12. To detect the acceptability level in KidneYou users.

Safety 13. To describe the safety profile in the two treatment groups.

Primary Endpoints

- To evaluate the achievement of a mean reduction of at least 10% of azoturia (g/24h) in Chronic Kidney Disease (CKD) KidneYou users exposed to a 3-month Nutritional Program (NP) compared to CKD KidneYou non-users exposed to the same 3-month NP.

OR

- To evaluate the achievement of a mean increase of at least 15% of distance (meters in the 6-MWT) in CKD KidneYou users exposed to a 3-month PA Program compared to CKD KidneYou non-users exposed to the same 3-month PA Program.

OR

- To evaluate the achievement of a mean decrease of at least 10% of perceived stress (according to the Perceived Stress Scale [PSS] of Cohen) in CKD KidneYou users exposed to a 3-month Mindfulness Program (MP) compared to CKD KidneYou nonusers and non-exposed to the same MP.

Safety Endpoint To assess the rate of adverse events, adverse device effects, abnormality of laboratory

Statistical Hypotheses This study is designed to test the null hypothesis that the percentage 'success' (intended as primary endpoint achievement) in KidneYou non-users is equal to the percentage 'success' in KidneYou users. The alternative hypothesis is that the percentage 'success' in KidneYou nonusers is different from the percentage 'success' in KidneYou users.

Sample Size Determination The sample size is estimated to provide statistical power for the primary endpoint. The sample size calculation is based on the combination of expected proportion of success in the control group and expected delta (Δ) of success in the experimental group.

With a significance level α equal to 0.05 and a power equal to 80%, a sample size of 190 subjects (95 per group) is required to detect as significant, if any, a success delta in favor of the experimental group equal to 20% (under the hypothesis of success rate of 40% in the control group and success rate of 60% in the experimental group).

Data Quality Assurance All participant data relating to the study will be recorded on eCRF unless transmitted to the sponsor or designee electronically (e.g., laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by electronically signing the eCRF.

The investigator must permit study-related monitoring, audits, Institutional Review Board/Ethic Committee review, and regulatory agency inspections and provide direct access to source data documents.

The sponsor or designee is responsible for the data management of this study including quality checking of the data.

Study monitors will perform ongoing source data verification to confirm that data entered into the eCRF by authorised site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH (International Conference on Harmonization) GCP (Good Clinical Practice), and all applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

- Age

1. Participant must be ≥18 years of age, at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
2. Participants with Chronic Kidney Disease (CKD) classified as Glomerular Filtration Rate (GFR) category G3b (30-44 ml/min/1.73 m2) or G4 (15-29 ml/min/1.73 m2); persistent albuminuria category A1 (<30 mg/g [<3 mg/mmol]) or A2 (30-300 mg/g [3-30 mg/mmol]); AND with presence of at least of the following causal etiologies: diabetes, arterial hypertension, chronic glomerulonephritis, cystic kidney diseases (e.g. polycystic kidney, nephronophthisis, cortical or tubular glomerular cysts, cystic diseases of the renal medulla, tuberous sclerosis, etc); AND with both abnormalities of kidney function (i.e., GFR and albuminuria) and structure (causal etiologies) present for >3 months, with implications for health.

   AND with a total score >12 in the Perceived Stress Scale (PSS) questionnaire by Cohen (Appendix E).

   Sex
3. Male and Female Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   Informed Consent
4. Capable of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

   - Other Criteria
5. Participants owning a mobile phone, willing to use mobile Apps and this type of technology (technology-savvy) and to download KidneYou.
6. Native speakers of Italian language or foreign subjects who have a full understanding of the Italian language, as the instructions and information for all health programs (i.e., dietary, physical activity, mindfulness) will only be given in Italian.

Exclusion Criteria:

- Medical Conditions

1. Any type of acute and/or chronic joint disease that prevents the patient from undergoing the recommended physical activities and interferes with the performance of the 6-MWT.
2. Any type of acute and/or chronic muscle diseases.
3. History or current evidence of depression, sleep disturbance, suicidal ideation or any mental (behavioural or psychological illness) disorder.
4. Patient's refusal or inability to follow dietary rules due to socio-economic or psychological distress.
5. Chewing disorder.
6. Lack of motivation to follow NP, PA program, psychological program and/or deterioration in the quality of life.
7. Positive hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody, Child-Pugh class C (Appendix G), at baseline visit.
8. Evidence to have tested positive for human immunodeficiency virus (HIV).
9. History or current evidence of drug or alcohol abuse.
10. History of QT prolongation and/or congenital long QT syndrome.
11. History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication are permitted.
12. Solid cancer, blood and/or hematopoietic cancer
13. Autoimmune diseases (i.e. systemic lupus erythematosus, scleroderma, rheumatoid arthritis, etc.).
14. Addison's disease.
15. Amyloidosis.

    - Prior/Concomitant Therapy
16. Any change (e.g., increase/decrease of medication dosage(s), termination of current medication(s), addition of new medication(s), replacement of one or more medication(s)) in the current patient's treatment strategy (concomitant therapies) due to subject's enrolment in this study.

    - Prior/Concurrent Clinical Study Experience
17. Participation in another clinical study with an Investigational Product administered in the last 6 months.

    - Diagnostic Assessments
18. Not applicable.

    - Other Exclusions
19. Involvement in the planning and/or conduct of the study (applies to both Advice Pharma S.r.l. staff and/or staff at the study site).
20. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
21. Previous enrolment or randomisation in the present study.
22. For women only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding.
23. As judged by the investigator, any evidence of CKD patient's condition which in the investigator's opinion makes it undesirable for the subject to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of changes in azoturia | Daily / Assessment at each month for three months
  The percentage of achievement of a mean reduction of at least 10 percent of azoturia (g/24h).
Evaluation of changes in distance covered | Daily / Assessment at each month for three months
  The achievement of a mean increase of at least 15 percent of distance (meters in the 6 Minutes Walking Test - 6MWT).
Evaluation of changes in Perceived Stress | Daily / Assessment at each month for three months
  The achievement of a mean decrease of at least 10 percent of perceived stress (according to the Perceived Stress scale of Cohen) in KidneyYou users exposed to a 3-month Nutritional Program, PA Program and Mindfulness Program compared to KidneyYou non-users and non-exposed to the same 3-month programs.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Flavio Ferri, Study Director — Advice Pharma Group S.r.l.
Locations (1):
- U.O. Nefrologia, Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Background] Cupisti A, Brunori G, Di Iorio BR, D'Alessandro C, Pasticci F, Cosola C, Bellizzi V, Bolasco P, Capitanini A, Fantuzzi AL, Gennari A, Piccoli GB, Quintaliani G, Salomone M, Sandrini M, Santoro D, Babini P, Fiaccadori E, Gambaro G, Garibotto G, Gregorini M, Mandreoli M, Minutolo R, Cancarini G, Conte G, Locatelli F, Gesualdo L. Nutritional treatment of advanced CKD: twenty consensus statements. J Nephrol. 2018 Aug;31(4):457-473. doi: 10.1007/s40620-018-0497-z. Epub 2018 May 24. PMID 29797247
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Johansen KL, Painter P. Exercise in individuals with CKD. Am J Kidney Dis. 2012 Jan;59(1):126-34. doi: 10.1053/j.ajkd.2011.10.008. Epub 2011 Nov 23. PMID 22113127
- [Background] Kang YS, Choi SY, Ryu E. The effectiveness of a stress coping program based on mindfulness meditation on the stress, anxiety, and depression experienced by nursing students in Korea. Nurse Educ Today. 2009 Jul;29(5):538-43. doi: 10.1016/j.nedt.2008.12.003. Epub 2009 Jan 13. PMID 19141364
- [Background] Huberty J, Green J, Glissmann C, Larkey L, Puzia M, Lee C. Efficacy of the Mindfulness Meditation Mobile App "Calm" to Reduce Stress Among College Students: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jun 25;7(6):e14273. doi: 10.2196/14273. PMID 31237569
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591